CLINICAL TRIAL: NCT06846034
Title: Effect of Acute Hypoxia on Renal Hemodynamic in Healthy Volunteers, Patients With Diabetes and Patients With Diabetes and Kidney Disease : Pilot Study.
Brief Title: Effect of Acute Hypoxia on Renal Hemodynamic in Healthy Volunteers, Patients With Diabetes and Patients With Diabetes and Kidney Disease
Acronym: DIAKIPOX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DIAKIPOX
Record Dates: First submitted 2025-02-13; First posted 2025-02-25 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Diabetes; Diabetic Kidney Disease; Hypoxia; Healthy Volunteer; Diabetic Nephropathies
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies; Hypoxia

STUDY DESIGN:
Intervention Model Description: It is a descriptive, prospective, open label, single centre, pilot study.
  This research aim to better understand the effect of hypoxia on intrarenal hemodynamic parameters of 3 groups :
  Group 1: Healthy volunteers Group 2: Patient with Type 2 Diabetes (DT2) without Diabetic Kidney Disease (DKD) Group 3: Patient with T2D and DKD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- acute hypoxia (Other): The participant will be exposed to 2 sequences : a 3-hour normoxia period and then a 2-hour hypoxia (FiO2=14.26% corresponding to 3000m altitude) period.
  Interventions: Other: Hypoxia administration study group; Combination Product: Renal clairance study

INTERVENTIONS:
Other: Hypoxia administration study group — Acute 2-hour hypoxia (14.5%FiO2 corresponding to 3000m altitude)
Combination Product: Renal clairance study — Assessment of renal clearance by measuring Glomerular Filtration Rate (GFR) after two agents infusion:
  * Aminohippurate Sodium (or or para-aminohippuric acid [PAH]) Inj 20% Diagnostic agent used to measure effective renal plasma flow (ERPF)
  * Iohexol Inj 300 MG/ML Diagnostic agent used to measure glomerular filtration rate (GFR)

SUMMARY:
Diabetes mellitus is a non-transmissible disease whose incidence is growing worldwide .

This pathology is defined by a chronic hyperglycaemia linked to a deficiency of either insulin secretion or its action or both. This increased prevalence is linked to the growing of the obese population on one hand, and to the ageing of the population, on the other hand, which is associated with an increased prevalence of metabolic diseases. The number of patients with diabetes, particularly type 2 diabetes (T2D) is regularly increasing. In France, the prevalence of diabetes is 4- 6% of the adult population.

Diabetic kidney disease (DKD) is a growing public health problem and therefore constitutes a major factor in progressive kidney disease. DKD has become the leading cause of end stage kidney disease (ESKD), requiring dialysis or transplantation.

Current routine screening for DKD is limited to detecting of impaired glomerular filtration rate (GFR) and/or elevated albuminuria, typically manifests in later stages of DKD. Therefore, the current methods to screen for DKD lack the resolution to capture the earliest functional changes associated with DKD.

Chronic renal hypoxia plays a crucial role in the development and progression of DKD and may affect Renal hemodynamic.

The aim to assess the feasibility of the measure of hypoxa-induced renal hemodynamics parameters.

ELIGIBILITY:
Inclusion Criteria:

For all participant :

1. No history of respiratory diseases
2. Affiliated person or beneficiary of the French social security scheme.
3. signed informed consent

Group 1 ( For healthy volunteers):

1. [18; 40] years old
2. No history of diabetes
3. No acute/long term > 3 months drug use except contraception
4. BMI: [18,5 - 29,9]kg/m2
5. eGFR > 60ml/min/1.73m2
6. Normal to midly increased albuminuria: defined as ACR < 3 mg/mmol

For all the patients with T2D (group 2 and 3):

1. Diagnosed T2D according to ADA criteria
2. [35; 75] years old
3. Stable treatment of diabetes and/or antihypertension for at least 2 months prior to inclusion
4. No proliferative diabetic retinopathy

Group 2 - For patients with T2D and no DKD:

* eGFR > 60ml/min/1.73m2 and
* Normal to midly increased albuminuria: defined as ACR < 3 mg/mmol

Group 3 - For patients with DKD:

* eGFR [45-60 ml/min/1.73m2] and/or
* Moderately to severely increased ACR ≥ 3 mg/mmol

Exclusion Criteria:

For all participants:

1. Active smoking
2. Contraindication to any of the agent (PAH, or iohexol or gadolinium) used in the study.
3. Contraindication to cardiac MRI, renal MRI, respiratory tests,
4. History acute coronary syndrome or coronary revascularization
5. Recent (<6 months) history of: Heart failure requiring hospitalisation or Stroke or transient ischemic neurologic disorder
6. Severe unstable hypertension (≥180 mmHg systolic or ≥110 mmHg diastolic blood pressure)
7. Resting oxygen saturation <95% at baseline
8. Any concomitant disease or condition that may interfere with the safety or the possibility for the patient to comply with or complete the study protocol.
9. History of severe mountain sickness (dizziness, headache, nausea/vomiting and incapaciting fatigue)
10. Consumption of SGLT2 inhibitors
11. Concurrent participation in another clinical research study
12. Pregnant or breastfeeding women, women of childbearing age who do not have effective contraception
13. Persons benefiting from enhanced protection under french national law
14. Persons under psychiatric care who are unable to give their consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Effective Renal Plasma Flow (ERPF) | 5 hours
  Measured by PAH clearance
Glomerular Filtration Rate | 5 hours
  Measured by Iohexol Clearance

SECONDARY OUTCOMES:
circulating and urinary mitochondrial metabolites | 8 days
  To investigate change of blood or urine metabolites : 2-ethyl 3-OH propionate, 3-hydroxy propionate, 3-hydroxy isovalerate, 3-methyl-crotonyl glycine, 3-hydroxy isobutyrate, Tiglyglycine, Aconitic acid, Citric acid, Glycolic acid, Homovanillic acid, Uracil, 3-methyl adipic acid.
blood pressure | 5 hours
  mean arterial pressure
heart rate | 5 hours
  heart rate
Lake Louise Questionnaire | 5 hours
  The Lake Louise Scoring was developed to assess the symptoms of acute mountain sickness in adults. It consist of 4 questions, each rated on a likert-type scale with 0-3 response options. Lower scores men a better outcome.
Oxygen saturation | 5 hours
  SpO2

OTHER OUTCOMES:
Renal Oxygenation Availability | 60 minutes
  Blood oxygen level dependent (BOLD) MRI
Cardiac Oxygenation Availability | 60 minutes
  Blood oxygen level dependent (BOLD) MRI

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Jean SAULNIER, MD PhD, Principal Investigator — CHU Poitiers
Locations (1):
- Centre Investigation Clinique CIC1402 - CHU Poitiers, Poitiers, France